CLINICAL TRIAL: NCT03570034
Title: Obalon Balloon System - Post-Approval Study
Brief Title: Obalon Balloon System Post-Approval Study
Acronym: PAS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Obalon Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-7500-0011
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Obalon Balloon System: Obalon Balloon System with moderate intensity Weight Loss Behavioral Modification Program
  Interventions: Device: Obalon Balloon System

INTERVENTIONS:
Device: Obalon Balloon System — Obalon Balloon System with a moderate intensity Weight Loss Behavioral Modification Program

SUMMARY:
The Obalon Balloon System - Post-Approval Study is a prospective, observational, and multi-center study.

DETAILED DESCRIPTION:
The Obalon PAS is a 1-year study that includes 6-month of Obalon Balloon therapy in conjunction of a weight loss behavior modification (WLBM) program and 6-month of continued WLBM program after balloon removal

ELIGIBILITY:
Inclusion Criteria:

* At least 22 years old
* BMI of 30-40 kg/m2

Exclusion Criteria:

* Contraindicated for the device
* Use of medications or medical devices known to induce weight gain or weight loss within the preceding 6 months.
* Known history of endocrine disorders affecting weight.
* Participation in any clinical study which could affect weight loss within the past year
* Known history or present condition of structural or functional disorders of the esophagus that may impede passage of the device through the gastrointestinal tract, including, Barrett's esophagus, esophagitis, dysphagia, achalasia, stricture/stenosis, esophageal varices, diverticula, or any other disorder of the esophagus
* Life expectancy less than 1 year or severe renal, hepatic, pulmonary or other medical condition, in the opinion of the investigator

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients aged 22 years and older, who are considered obesity Class I or II with a BMI of 30.0-40.0 kg/m2; and, have failed to lose weight through diet and exercise
  * Patients willing to commercially purchase the device.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-09-13 (Estimated); Study Completion 2021-03-13 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Event | 6-Month
  Device or Procedure related Serious Adverse Event
Percentage of Patients with at least 5% TBWL | 6-Month
  Percentage of Patients with at least 5% TBWL
Mean % TBWL | 6-Month
  Mean %TBWL

CONTACTS AND LOCATIONS:
Overall Officials: Shelby Sullivan, MD, FACG, Principal Investigator — University of Colorado, Denver; Rachel Moore, MD, FACS, FASMBS, Principal Investigator — Surgical Specialist of Louisiana
Locations (15):
- United States (15):
  - Smart Dimensions Weight Loss, Fountain Valley, California
  - Davtyan Medical Weight Loss and Wellness, Glendale, California
  - Lifetime Surgical Weight Loss, Los Gatos, California
  - SkyLex Health, Santa Monica, California
  - University of Colorado Denver, Aurora, Colorado
  - Surgical Specialists of Louisiana, Metairie, Louisiana
  - New Jersey Bariatric Center, Springfield, New Jersey
  - Greenwich Village Gastroenterology, Poughkeepsie, New York
  - New York Bariatric Group, Roslyn Heights, New York
  - JourneyLite Physicians, Cincinnati, Ohio
  - Artisan Cosmetic Surgery, Toledo, Ohio
  - Minimally Invasive Surgical Associates, Dallas, Texas
  - Snow Bariatic Center, Flower Mound, Texas
  - Ultimate Bariatrics, Fort Worth, Texas
  - Bariatric Medical Institute of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No